CLINICAL TRIAL: NCT03038555
Title: The Study of Prevention and Intervention Strategy of Gestational Diseases Based on Cohort
Brief Title: China Obstetrics Alliance Cohort Study
Acronym: COACS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: The Third Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Obstetrics & Gynecology Hospital of Fudan University (Other); Tongji Medical College of Huazhong University of Science & Technology (Unknown); Xinjiang Maternity & Children Health Care Hospital (Unknown); Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Dunjin Chen, Guangzhou Institute of Obstetrics & Gynecology, The Third Affiliated Hospital of Guangzhou Medical University
Other Study IDs: 2016YFC1000405
Record Dates: First submitted 2017-01-26; First posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Preeclampsia
Keywords: Medical staff; preeclampsia; cohort study; further effect
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Store the blood samples (serum, blood and plasma) of both the experimental group and control group and their children.
  These additional samples were be centrifuged and treated and stored in a collection of biological samples of total serum and plasma and blood at the Biobank of The Third Affiliated Hospital of Guangzhou Medical University at -80 ° C

GROUPS / COHORTS (2):
- Disease group (subject to strategy): Choose subjects that have ever got PE before as the diseases group.
- Control group: Pair the same age, gestational weeks, children's gender and healthy subject as a control group in the ratio of 1:1. The control group should exclude subject that have ever got heart or lung diseases, diabetes, chronic nephrosis, immune disease and other hereditary disease.

SUMMARY:
Preeclampsia (PE) is one of a common type of hypertensive disorder complicating pregnancy (HDCP). It is a class of clinical syndromes which shows relevant symptoms, hypertension and proteinuria after 20 weeks pregnant as main characteristic, and may accompany with fetal anomaly and systemic multi-system organs damage. Several complications, such as eclamptic seizures, coma, intracranial hemorrhage (ICH), cardiac failure, pneumonedema, hepatic failure, kidney failure, placental abruption and disseminated intravascular coagulation (DIC), may be threat to the life of the mother as well as fetal. Thus, the disease is one of the core issues that cause the maternal and perinatal death. Morbidity of PE is approximately 3% to 5%. Morbidity has significant differences between different populations. According to the data, from 1995 to 2004, HDCP morbidity in four hospitals in Guangzhou was 5.78%, and in the HDCP, mild preeclampsia and severe preeclampsia were accounted for 72.22% and 27.78% respectively. Meanwhile, HDCP morbidity decreased from 9.4% (1984 to 1989) to 5.57% (1989 to 1998).

In 1996, the American Congress of Obstetricians and Gynecologists (ACOG) gave new classification of HDCP based on the characteristic of disease symptoms, divide into five groups; gestational hypertension, preeclampsia, eclampsia, chronic hypertension complicated with preeclampsia and chronic hypertension. The pathogenesis of PE remains unclear so far. The frequent sight is that PE caused by multiple reactions by a number of factors affect. Physiologically, mainly altered of PE is increased blood viscosity and systemic vascular spasm which cause hypoxic-ischemic of multiple key organs, such as the placenta, kidney, liver and brain. The research theory includes abnormal trophoblast invasion, immune response abnormal or increase, genetic susceptibility, coagulation disorders or thrombophilia, abnormal angiogenesis, endothelial cell damage, abnormal levels of carbonic oxide, increase of oxygen radical, abnormal metabolism of calcium ion, heterotrophia and so on. However, there are numbers of epidemiologic study have analyzed high risk factor of PE which provides significant medical evidence of prevention, early diagnosis and early treatment for PE, there is only little study focus on susceptibility gene and pathogenic genetic variation. Nowadays, there are numerous clinical phenotype are considered to exist, different phenotype gives different inheritance and epigenetics. Thus, our group will examine the onset of type and characteristics of PE by a retrospective cohort study to discuss if susceptibility gene and pathogenic genetic variation were existing in PE patients, also to find the relativity between clinical phenotype and genotype. Moreover, this study is trying to reach the effect of PE on the patients' health as well as their children. Thus, can predict the health status of PE patients and their children, and so can prevent (avoid or delay) of the patients from late complications and disease in their children.

DETAILED DESCRIPTION:
1. All female staff that works, examination and delivery in the Third Affiliated Hospital of Guangzhou Medical University from Dec 1995 to Dec 2016 should be in the cohort. Collect all information; include clinical examination and medical examination, science the subject work in the hospital. Collect the perinatal data; include obstetric information, past medical history, family history and so on. Build the database and analyze the relative factor.
2. From all subjects, choose subjects that have got PE before as the experimental group. Pair the same age, gestational weeks, children's gender and healthy subject as a control group in the ratio of 1:1. The control group should exclude subject that have ever got heart or lung diseases, diabetes, chronic nephrosis, immune disease and other hereditary disease. Store the blood samples (serum, blood and plasma) of both the experimental group and control group and their children. Compare the differences of functional parameter between two groups both before and after delivery, which include blood pressure, blood glucose and blood lipids. Moreover, compare the function of heart, liver and kidney and genetic material (DNA and RNA).
3. Diagnostic standard of PE refer to People's Medical Publishing House <Obstetrics and Gynecology> 8th edition. Confirm the diagnostic standard of HDCP and relative disease include PE will make sure the veracity and uniformity of diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Choose subjects that have got PE before as the experimental group. Pair the same age, gestational weeks, children's gender and healthy subject as a control group in the ratio of 1:1.

Exclusion Criteria:

* Subject that have ever got heart or lung diseases, diabetes, chronic nephrosis, immune disease and other hereditary disease.

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Choose subjects that have got PE before as the experimental group. Pair the same age, gestational weeks, children's gender and healthy subject as a control group in the ratio of 1:1. The control group should exclude subject that have ever got heart or lung diseases, diabetes, chronic nephrosis, immune disease and other hereditary disease.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
track the difference between preeclampsia and normal | 2 years
  Our main judgement criterion allowing to distinguish patients with preeclampsia from those without disease

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Guangzhou Institute of Obstetrics & Gynecology, Guangzhou, Guangdong
  - Tongji Medical College Huazhong University of Science & Technology, Wuhan, Hubei
  - Shandong Provincial Hospital, Jinan, Shandong
  - Xinjiang Maternity & Children Health Care Hospital, Ürümqi, Xinjiang
  - Obstetrics and Gynecology Hospital of Fudan University, Shanghai